CLINICAL TRIAL: NCT02448979
Title: Randomized Control Study on Surgical Treatment for Middle and Lower Thoracic Esophageal Cancer Patients Without Upper Mediastinal Lymph Node Metastasis Through Left Versus Right Transthoracic Approach
Brief Title: Esophagectomy in Middle and Lower Thoracic Esophageal Cancer Patients Through Left Versus Right Transthoracic Approach
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Henan Cancer Hospital (Other Government); Hebei Medical University Fourth Hospital (Other); Harbin Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Hunan Cancer Hospital (Other); Sun Yat-sen University (Other); Zhejiang Cancer Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jie He, President, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKTRDP-2015BAI12B08-01
Record Dates: First submitted 2015-05-08; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left thoracotomy (Active Comparator): Esophagectomy through left side transthoracic approach, with esophagogastric anastomosis above aortic arch and two-field lymphadenectomy (thoracic and abdominal lymph node)
  Interventions: Procedure: Left thoracotomy
- Right thoracotomy (Active Comparator): Esophagectomy through right side transthoracic approach, with esophagogastric anastomosis above azygos vain arch or on the top of chest cavity and two-field lymphadenectomy (thoracic and abdominal lymph node)
  Interventions: Procedure: Right thoracotomy

INTERVENTIONS:
Procedure: Left thoracotomy — Transthoracic approach is the surgical procedure including the open and minimally invasive thoracotomy.
  Arms: Left thoracotomy
Procedure: Right thoracotomy — Transthoracic approach is the surgical procedure including the open and minimally invasive thoracotomy.
  Arms: Right thoracotomy

SUMMARY:
Esophageal carcinoma is an aggressive malignant disease with poor prognosis. Surgical resection remains the most effective method for this malignancy. Although different approaches have been studied for the surgical resection of thoracic esophageal cancer, little evidence has been achieved due to lack of large scale multicenter randomized trials with regard to this issue: whether left transthoracic approach or right transthoracic approach is the optimal surgical approach for treating middle and lower thoracic esophageal cancer without upper mediastinal lymph node metastasis. The purpose of this study is to compare the postoperative local recurrence rate and long-term outcome of esophagectomy through left and right transthoracic approach in the middle and lower thoracic esophageal cancer patients without preoperative upper mediastinal lymph node metastasis.

DETAILED DESCRIPTION:
Esophageal carcinoma is an aggressive malignant disease with poor prognosis. Surgical resection remains the most effective method for this malignancy. As to the middle and lower thoracic esophageal cancer patients without upper mediastinal lymph node metastasis, the rational transthoracic approach either through right or left chest has not been clarified to date due to lack of large scale multicenter randomized trials. Although some randomized trials had been finished in single-center, there is no enough evidences that all lower and middle thoracic esophageal cancer patients should be surgically treated throuhg right chest approch. It is widely recognized that left thoracotomy approach(Sweet procedure) is not appropriate in the patients with upper mediastinal lymph node metastasis, because patients can benefit from the right thoracotomy approach, through which upper mediastinal lymph node can be dissected completely and may get a better long-term survival.Therefore,in this study, the enrolled patients are the middle and lower thoracic esophageal cancer patients without preoperative upper mediastinal lymph node metastasis by CT and/or ultrasound, and 10 hospitals will participate this study. Through comparison in postoperative complications and long term outcomes as well as locoregional recurrence between the left and right apppoach, hopefully we can answer the question whether the right or left transthoracic procedure is the optimal approach for treating middle and lower thoracic esophageal cancer patients without preoperative upper mediastinal lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proved squamous cell esophageal cancer without any previous anti-tumor therapy;
2. The preoperative clinical TNM stage: cT1b-3N0-1M0;
3. Adequate function of heart, lung, liver, brain and kidney, which can tolerate esophagectomy either through left or right thoracotomy;
4. Without any preoperative distant metastases confirmed by preoperative examination such as chest and abdominal CT, brain MRI and bone scan or PET-CT;
5. No evidence showing suspicious upper mediastinal lymph node metastasis (short diameter of LN <0.8cm or shortest diameter / longest diameter <0.65) by the thoracic and abdominal CT and endoscopic ultrasonography(EUS).
6. Willing to participate the clinical trial and sign informed consent before being enrolled into clinical trail.

Exclusion Criteria:

1. Non-squamous cell esophageal carcinoma or has any previous anti-cancer therapy before surgery;
2. The preoperative clinical TNM stage reaches: N2-3 or M1;
3. Inadequate cardiopulmonary, liver, brain and kidney function for tolerating the esophagectomy ;
4. Previous history of malignancy;
5. Unwilling to participate the clinical trial and refuse to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Long term survival | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years
Degree of lymph node dissection | 3 years
Postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mao YS, Gao SG, Li Y, Hao AL, Liu JF, Li XF, Rong TH, Fu JH, Ma JQ, Xu MQ, Zhang RQ, Xiao GM, Fu XN, Chen KN, Mao WM, Liu YY, Liu HX, Zhang ZR, Fang Y, Fu DH, Wei XD, Yuan LG, Muhammad S, Wei WQ, Chiu PW, Lloyd S, Schlottmann F, Meredith K, Pimiento JM, Gao YB, He J. Efficacy and safety of esophagectomy via left thoracic approach versus via right thoracic approach for middle and lower thoracic esophageal cancer: a multicenter randomized clinical trial (NST1501). Ann Transl Med. 2022 Aug;10(16):904. doi: 10.21037/atm-22-3810. PMID 36111056